CLINICAL TRIAL: NCT02443064
Title: Pharmacokinetics/ Pharmacodynamics (PK/PD) Study of Vancomycin in the Treatment of Methicillin-resistant Staphylococcus Aureus（MRSA） Blood Stream Infection (Septicemia) and Endocarditis in Chinese Patients
Brief Title: Pharmacokinetics/ Pharmacodynamics (PK/PD) Study of Vancomycin
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang University (Other)
Collaborators: Shengjing Hospital (Other); Tianjin Medical University Cancer Institute and Hospital (Other); Qilu Hospital of Shandong University (Other); First Affiliated Hospital, Sun Yat-Sen University (Other); Guangzhou General Hospital of Guangzhou Military Command (Other); The First Affiliated Hospital of Soochow University (Other); The First Affiliated Hospital with Nanjing Medical University (Other); Zhejiang Provincial Hospital of TCM (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Principal Investigator, Yong-Hong Xiao, Vice Director, China State Key Laboratory for Diagnosis and Treatment of Infectious Diseases, the First Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou., Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XYH-88; zju-vancamycin (Other: zju-vancamycin)
Record Dates: First submitted 2014-11-23; First posted 2015-05-13 (Estimated); Last update posted 2015-05-13 (Estimated); Status verified 2015-05

CONDITIONS: Blood Stream Infections; Endocarditis; MRSA
Keywords: Pharmacokinetics/pharmacodynamics; vancomycin; blood stream infections; Chinese patients; MRSA
MeSH Terms: conditions — Endocarditis | interventions — Vancomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MRSA blood stream infection patient (Experimental): Intervention:Vancomycin
  Dosing:
  15-20mg/kg, IV,q 12~8h (or 1 g, IV, q12~8h) for adult patient with normal renal function; Dosage should be adjusted by blood creatinine clearance in patients with impaired renal function; Administration route： 1~2 h/ dosing, IV
  Drug combination:
  Drug combination is not recommended for patients with simple MRSA infection; Rifampicin can be combined in case of MRSA artificial valve endocarditis; Anti-G- antibacterial agents can be combined in case of concurrent G- bacterial infections.
  Duration:
  Septicemia: 2~4 weeks Endocarditis: 6~8 weeks
  Interventions: Drug: Vancomycin

INTERVENTIONS:
Drug: Vancomycin — Vancomycin was administered for Chinese patients with MRSA blood stream infection and endocarditis Pharmacokinetics: 5 blood samples collected at steady state for the determination of plasma concentrations for population pharmacokinetics (PPK) analysis.
  Microbiology: blood cultures for MRSA isolation, MIC of vancomycin against MRSA; molecular typing will be analyzed on bacterial strains including heterogeneous vancomycin-intermediate Staphylococcus aureus (hVISA) and vancomycin-intermediate Staphylococcus aureus （VISA); Safety evaluation: hepatic and renal function, blood routine test, and so on.

SUMMARY:
1. Drug resistance of G+ cocci is a severe healthcare problem. According to the Ministry of Health National Antimicrobial Resistant Investigation Net (mohnarin) surveillance report, the isolation rate of MRSA is some 60% in China. MRSA infection has become a serious clinical problem;
2. Vancomycin is a bactericidal glycopeptide antibiotic which inhibits bacterial growth by hindering the synthesis of cell wall in bacteria. It exerts strong antibiotic effect to Gram+ bacteria. It is indicated for serious staphylococcus infections especially MRSA infection and has become the gold standard agent in MRSA treatment;
3. Vancomycin is a time-dependent antibiotic, its clinical and microbiological efficacy is related to area under curve（ AUC）/minimum inhibitory concentration （MIC ）(AUIC). Cmin at steady state is an surrogate parameter of AUIC, which is closely associated to the efficacy;
4. AUIC >400 and Cmin between 15~20 mg/L are recommended for effective vancomycin treatment by Infectious Diseases Society of America （IDSA） although it is still disputable;
5. Due to the absence of PK/PD study on vancomycin in China, administration of vancomycin is performed in reference to the recommendation of IDSA. Its suitability to Chinese patients is still to be clarified;
6. Plasma concentrations of vancomycin vary significantly between population and individuals. Factors such as large-volume fluid infusion, hypoproteinemia and renal clearance, etc. will influence the distribution and excretion of vancomycin, resulting in different plasma concentrations between individuals. Results of PK studies differ greatly between China and abroad. Administration based on the AUIC or Cmin recommended by IDSA would not be suitable to Chinese patients. Given the definite long-term benefit of vancomycin treatment, the AUIC or Cmin suitable to Chinese patients must be identified by clinical study.
7. The PK/PD study on vancomycin in the treatment to MRSA septicemia and endocarditis is of great significance for more reasonable use and improved therapeutic efficacy of MRSA infection.

DETAILED DESCRIPTION:
Study design:

A multi-center, non-controlled, open-labeled observational study

Research objectives

Primary objective:

To explore the PK/PD target value (AUIC) of vancomycin in the treatment of MRSA septicemia and endocarditis in Chinese patients.

Secondary objective:

To detect the therapeutic efficacy and safety of vancomycin in the treatment of MRSA septicemia and endocarditis in Chinese patients.

To exam the relationship between the Cmin of vancomycin and its efficacy in the treatment to MRSA septicemia and endocarditis.

To explore the relationship between MRSA molecular type and vancomycin therapeutic efficacy

Medicine and administration

Drug:

Vancomycin

Dosing:

15~20 mg/kg, IV, q 12~8h (or 1 g, IV, q12~8h) for adult patient with normal renal function; Dosage should be adjusted by blood creatinine clearance in patients with impaired renal function; Administration route： 1~2 h/ dosing, IV

Drug combination:

Drug combination is not recommended for patients with simple MRSA infection; Rifampicin can be combined in case of MRSA artificial valve endocarditis; Anti-G- antibacterial agents can be combined in case of concurrent G- bacterial infections.

Duration:

Septicemia: 2~4 weeks Endocarditis: 6~8 weeks

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years, male or female;
2. diagnosed as MRSA septicemia or endocarditis; Septicemia clinical manifestations of infection; MRSA infection confirmed by blood culture; Endocarditis: diagnosed according to modified Duke Criteria
3. no therapy with effective anti-MRSA drugs 72 hours prior to the study; Effective anti-MRSA drugs used in China include: vancomycin, norvancomycin, teicoplanin, linezolid, daptomycin, tigecycline, and fusidic acid.

Exclusion Criteria:

1. those being allergic to glycopeptides antibiotics;
2. those with osteomyelitis, central nervous system infection or other septic migrations (except for endocarditis);
3. patients with catheter-related bloodstream infection who cannot withdraw catheter;
4. those during chemotherapy for cancer or leukemia;
5. those with agranulocytosis;
6. those with HIV infection;
7. women in pregnancy or lactation;
8. patients receiving vancomycin for less than 72 hours;
9. patients participating in any other clinical trial in 3 months prior to the study (not limited to trials for antibiotics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-01; Primary Completion 2016-01 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
AUC/MIC of vancomycin in each patient | Participants will be followed for the duration of hospital stay, an expected average of 4 weeks

SECONDARY OUTCOMES:
Number of participants with negative blood culture at the end of treatment | Participants will be followed during vancomycin treatment and in average of 4 weeks after vancomycin treatment
Number of participants with adverse events | Participants will be followed during vancomycin treatment and in average of 4 weeks after vancomycin treatment
Number of participants survival | Participants will be followed during vancomycin treatment and in average of 4 weeks after vancomycin treatment

CONTACTS AND LOCATIONS:
Overall Officials: Yong-hong Xiao, MD, Principal Investigator — The First Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, China
Locations (1):
- Yong-Hong Xiao, Hangzhou, Zhejiang, China

REFERENCES:
- [Background] Kullar R, Davis SL, Levine DP, Rybak MJ. Impact of vancomycin exposure on outcomes in patients with methicillin-resistant Staphylococcus aureus bacteremia: support for consensus guidelines suggested targets. Clin Infect Dis. 2011 Apr 15;52(8):975-81. doi: 10.1093/cid/cir124. PMID 21460309
- [Background] Brown J, Brown K, Forrest A. Vancomycin AUC24/MIC ratio in patients with complicated bacteremia and infective endocarditis due to methicillin-resistant Staphylococcus aureus and its association with attributable mortality during hospitalization. Antimicrob Agents Chemother. 2012 Feb;56(2):634-8. doi: 10.1128/AAC.05609-11. Epub 2011 Nov 28. PMID 22123681
- [Background] Liu C, Bayer A, Cosgrove SE, Daum RS, Fridkin SK, Gorwitz RJ, Kaplan SL, Karchmer AW, Levine DP, Murray BE, J Rybak M, Talan DA, Chambers HF; Infectious Diseases Society of America. Clinical practice guidelines by the infectious diseases society of america for the treatment of methicillin-resistant Staphylococcus aureus infections in adults and children. Clin Infect Dis. 2011 Feb 1;52(3):e18-55. doi: 10.1093/cid/ciq146. Epub 2011 Jan 4. PMID 21208910
- [Background] Anonymous. Expert consensus on the use of vancomycin(2011). Chin J of New Drug & Regimen. 2011，30（8）：561-56
- [Result] 1.Xiao YH, et al. 2010 report of Mohnarin. Chin J Nosocomial Infect. 2012, 22(22):4946-4952
- [Result] Moise-Broder PA, Forrest A, Birmingham MC, Schentag JJ. Pharmacodynamics of vancomycin and other antimicrobials in patients with Staphylococcus aureus lower respiratory tract infections. Clin Pharmacokinet. 2004;43(13):925-42. doi: 10.2165/00003088-200443130-00005. PMID 15509186